CLINICAL TRIAL: NCT02722343
Title: Phase I Exploratory Pharmacodynamic Study of Tenofovir-Based Products
Brief Title: Exploratory Pharmacodynamic Study of Tenofovir-Based Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: Eastern Virginia Medical School (Other); University of North Carolina (Other); Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A15-140
Record Dates: First submitted 2016-03-09; First posted 2016-03-30 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: HIV
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir intravaginal ring (Experimental): The tenofovir intravaginal ring (TFV IVR) is 55.0 mm in diameter, consisting of a single segment of polyurethane tubing with an outer diameter of 5.5 mm and filled with white TFV-containing paste. The IVR delivers 8-10mg/day of TFV.
  Interventions: Drug: Tenofovir intravaginal ring
- Truvada oral tablets (Active Comparator): The tablets contain 200mg emtricitabine combined with 300mg tenofovir disoproxil fumarate (300mg). The tablets are commercially available as Truvada. The tablets are blue, capsule-shaped, film-coated, debossed with "GILEAD" on one side and with "701" on the other side
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Tenofovir intravaginal ring — The participant will wear the intravaginal ring consecutively for 14 days and nights. Following study product use and at study visit 4, blood and genital tract samples will be taken (to include cervico-vaginal fluid and tissue)
  Other Names: Tenofovir disoproxil fumarate intravaginal ring; TFV IVR
  Arms: Tenofovir intravaginal ring
Drug: Truvada — The participant will take the tablet for 14 days. taking one tablet each morning. Following study product use and at study visit 4, blood and genital tract samples will be taken (to include cervico-vaginal fluid and tissue)
  Other Names: Emtricitabine/tenofovir disoproxil fumarate tablets
  Arms: Truvada oral tablets

SUMMARY:
This single site study is designed to describe and measure the efficacy of oral versus vaginal dosing of TFV-based products, specifically emtricitabine/tenofovir disoproxil fumarate oral tablets (Truvada) vs tenofovir intravaginal rings (IVR).

DETAILED DESCRIPTION:
This study will compare an investigational intravaginal ring containing tenofovir (TFV) with an FDA approved medication in tablet form called Truvada®. It will assess and compare the ability of the tablet and intravaginal ring to prevent HIV transmission (human immunodeficiency virus, the virus that causes AIDS).

The study will enroll healthy, non-pregnant, HIV negative, premenopausal women (aged 18-50, with regular menstrual cycles) who are not at risk of pregnancy.

The enrollment goal is for 20 participants to complete the study.

Participants will be assigned to use one of the study products: oral tablet or intravaginal ring. Participants will take the oral tablet each day for 14 days or wear the intravaginal ring all day and night for 14 days/nights. Blood, genital fluid samples and genital tissue samples (biopsies) will be taken at two visits. These sample collections will take place before and after use of the assigned study product. The samples will be tested to:

1. Determine the levels of drug in the blood and genital tissue samples
2. See if the samples taken from the vagina and cervix after use of study product, provides protection from HIV in the laboratory
3. Ensure that the laboratory test used to measure HIV infection in the samples performs well when used repeatedly.

In addition this study will also evaluate the returned TFV rings to see whether they were used as instructed.

ELIGIBILITY:
Inclusion Criteria:

* General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes) and with an intact gastrointestinal tract, uterus and cervix
* Currently have regular menstrual cycles of 21-35 days by participant record
* Willing to abstain from vaginal intercourse and any other vaginal activity including use of vaginal products (tampons, spermicides, lubricants, and douches) other than study products:

  * 48 hours before Visit 2 until six days after Visit 2
  * 48 hours before Visit 3 until six days after Visit 4
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection
* Estimated calculated creatinine clearance (eCcr) of at least 60 mL/min
* History of Pap smears and follow-up consistent with standard clinical practice as outlined in the study manual or willing to undergo a Pap smear at Visit 1
* Protected from pregnancy by one of the following:

  * sterilization of either partner
  * abstinence
  * same sex relationship
  * condoms
  * combined contraceptives (including oral, patch)
  * copper IUD
* Willing and able to comply with protocol requirements including swallowing tablets
* Willing to give voluntary consent and sign an informed consent form

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant or within two calendar months from the last pregnancy outcome. Note: if recently pregnant must have had at least two spontaneous menses since pregnancy outcome
* Injection of Depo-Provera in the last 10 months or use of other progestin-only based contraceptive (including hormonal IUD)
* Currently breastfeeding or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study products, topical anesthetic, or to both silver nitrate and Monsel's solution
* In the last three months, diagnosed with or treated for any STI, by self report
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, HIV, or Hepatitis B surface antigen (HBsAg) Note: Women with a history of genital herpes who have been asymptomatic for at least three months may be considered for eligibility
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, or antivirals (e.g., acyclovir, valacyclovir, Viread®, Atripla®, Emtriva®, or Complera®)
* Current or anticipated chronic use of NSAIDS, or Tylenol for the duration of the study
* Grade 2 or higher laboratory abnormality, per the 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data
* Known current drug or alcohol abuse which could impact study compliance
* Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
p24 antigen production in cervico-vaginal tissues infected with HIV | Day 14
  • Assess p24 antigen production in cervicovaginal tissues infected ex vivo with HIV-1BaL at baseline and after using Truvada tablets or tenofovir intravaginal ring
Analysis of integrated DNA | Day 14
  Integrated viral DNA in cervicovaginal tissues infected ex vivo with HIV-1BaL at baseline and after using Truvada tablets or tenofovir intravaginal ring
Anti-HIV activity in cervicovaginal fluid (CVF) | Day 14
  Anti-HIV activity in cervicovaginal fluid at baseline and after using Truvada tablets and tenofovir intravaginal ring

SECONDARY OUTCOMES:
Cervicovaginal tissue, fluid and plasma concentrations of tenofovir | Day 14
  Concentrations after use of Truvada tablets and tenofovir intravaginal ring
Cervicovaginal tissue concentration of tenofovir diphosphate | Day 14
  Concentrations after use of Truvada tablets and tenofovir intravaginal ring.
Cervicovaginal tissue, fluid and plasma concentrations of emtricitabine | Day 14
  Concentrations after use of Truvada tablets and tenofovir intravaginal ring.
Cervicovaginal tissue concentration of emtricitabine triphosphate | Day 14
  Concentrations after use of Truvada tablets and tenofovir intravaginal ring.
Endogenous nucleotide concentrations in cervicovaginal tissue | Day 14
  Endogenous nucleotides; dATP and dCTP concentrations in cervicovaginal tissue after use of Truvada tablets and tenofovir intravaginal ring

OTHER OUTCOMES:
Adherence markers in used IVRs | Day 14
  Adherence biomarkers from used IVRs returned to clinic after two weeks of use

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Thurman, M.D., Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ouattara LA, Thurman AR, Jacot TA, Cottrell M, Sykes C, Blake K, Fang X, Ju S, Vann NC, Schwartz J, Doncel GF. Genital Mucosal Drug Concentrations and anti-HIV Activity in Tenofovir-Based PrEP Products: Intravaginal Ring vs. Oral Administration. J Acquir Immune Defic Syndr. 2022 Jan 1;89(1):87-97. doi: 10.1097/QAI.0000000000002820. PMID 34878438